CLINICAL TRIAL: NCT01542684
Title: Phase II Study of Azacytidine Followed by GM-CSF in Patients With Low- or Intermediate-1- Risk Myelodysplastic Syndrome (MDS)
Brief Title: Study of Azacytidine Followed by GM-CSF in Patients With Myelodysplastic Syndrome (MDS)
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Slow Accrual
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2011-1123
Record Dates: First submitted 2012-02-27; First posted 2012-03-02 (Estimated); Results first posted 2014-04-30 (Estimated); Last update posted 2014-04-30 (Estimated); Status verified 2014-03

CONDITIONS: Leukemia
Keywords: Leukemia; Myelodysplastic Syndrome; MDS; Azacytidine; 5-Azacytidine; 5-AZA; Vidaza; 5-AZC; Aza-CR; Ladakamycin; NSC-102816; GM-CSF; Sargramostim; Leukine
MeSH Terms: conditions — Leukemia; Myelodysplastic Syndromes | interventions — Azacitidine; Granulocyte-Macrophage Colony-Stimulating Factor; sargramostim

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Azacytidine + GM-CSF (Experimental): Azacytidine administered intravenously (IV) or subcutaneously (SQ) at starting dose of 40 mg/m^2, daily for 4 days.
  GM-CSF administered IV or subcutaneously at 250 mcg/m^2 one day (the next day) after completion of azacytidine treatment, for 3 consecutive days.
  Each treatment cycle will last at least 4 weeks
  Interventions: Drug: Azacytidine; Drug: GM-CSF

INTERVENTIONS:
Drug: Azacytidine — Starting dose: 40 mg/m^2 intravenously (IV) or subcutaneously (SQ) daily for 4 days.
  Other Names: 5-Azacytidine; 5-AZA; Vidaza; 5-AZC; AZA-CR; Ladakamycin; NSC-102816
Drug: GM-CSF — 250 mcg/m^2 IV or SQ one day (the next day) after completion of azacytidine treatment, for 3 consecutive days.
  Other Names: Saragramostim; Leukine

SUMMARY:
The goal of this clinical research study is to learn if the combination of azacitidine and GM-CSF can help to control MDS. The safety of these drugs will also be studied.

Azacitidine is designed to block certain proteins that stop the function of tumor-fighting genes. By blocking the "bad" proteins, the tumor-fighting genes may be able to work better.

Granulocyte-macrophage colony-stimulating factor (GM-CSF) is designed to help produce white blood cells. This may help to fight infections.

DETAILED DESCRIPTION:
Study Drug Administration:

If you are found to be eligible to take part in this study, on Days 1-4 of every cycle, you will receive azacitidine by vein over 15-30 minutes.

You may receive drugs to help prevent nausea and vomiting before you receive your dose of azacitidine.

On Days 5-7 of every cycle, you will receive GM-CSF by vein over about 15 minutes or by injection.

Each study cycle will be about 4-6 weeks, depending on the study doctor's decision.

Study Visits:

One (1) time each week during every cycle, blood (about 2-3 teaspoons) will be drawn for routine tests.

At any time, if your doctor thinks it is needed, you will have a bone marrow aspirate to check the status of the disease.

Length of Study:

You may continue taking the study drugs for as long as the doctor thinks it is in your best interest. You will no longer be able to take the study drugs if the disease gets worse, if intolerable side effects occur, or if you are unable to follow study directions.

Your follow-up visits will be per standard of care for the disease.

This is an investigational study. Both azacitidine and GM-CSF are FDA approved and commercially available for the treatment of MDS. The study drug combination to treat MDS is considered investigational.

Up to 40 patients will take part in this study. All will be enrolled at MD Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with low- or intermediate-1-risk MDS according to the International Prognostic Scoring System (IPSS) classification
2. Signed informed consent indicating that patients are aware of the investigational nature of this study in keeping with the policies of UT MD Anderson Cancer Center.
3. Age >/= 18 years old.
4. Prior therapy with growth factor support, lenalidomide, or other investigational agents is allowed.
5. Previously untreated patients are eligible for this study.

Exclusion Criteria:

1. Any previous adverse reaction (>/= Common Terminology Criteria for Adverse Events (CTCAE) grade 2) to GM-CSF.
2. Prior treatment with azacytidine or decitabine.
3. Unresolved diarrhea >/= CTCAE grade 2.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2012-03; Primary Completion 2013-04 (Actual); Study Completion 2013-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Zeev Estrov, MD, Principal Investigator — UT MD Anderson Cancer Center
Locations (1):
- UT MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: UT MD Anderson Cancer Center Website — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment Period: 3/15/2012 through 1/14/2013. All participants recruited at The University of Texas MD Anderson Cancer Center.
Groups:
- Azacytidine + GM-CSF: Azacytidine administered intravenously (IV) or subcutaneously (SQ) at starting dose of 40 mg/m^2, daily for 4 days.
  Granulocyte-macrophage colony-stimulating factor (GM-CSF) administered IV or subcutaneously at 250 mcg/m^2 one day (the next day) after completion of azacytidine treatment, for 3 consecutive days.
  Each treatment cycle lasts at least 4 weeks.
Period: Overall Study
Arm/Group | Azacytidine + GM-CSF
Started | 8
Completed | 8
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Azacytidine + GM-CSF: Azacytidine administered intravenously (IV) or subcutaneously (SQ) at starting dose of 40 mg/m^2, daily for 4 days.
  GM-CSF administered IV or subcutaneously at 250 mcg/m^2 one day (the next day) after completion of azacytidine treatment, for 3 consecutive days.
  Each treatment cycle lasts at least 4 weeks.
Arm/Group | Azacytidine + GM-CSF
Number analyzed (Participants) | 8
Age, Continuous [Median (Full Range); unit: Years] | 69 [54 to 82]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 7
Region of Enrollment [Number; unit: participants]
  United States | 8

OUTCOME MEASURES:

1. Primary Outcome: Overall Response Rate (ORR)
Description: ORR is percentage total participants with overall response (Complete Response (CR) or Partial Response (PR)) within two treatment cycles. Response based on modified International Working Group (IWG) criteria: Complete response - Bone marrow: 5% myeloblasts with normal maturation of all cell lines, Persistent dysplasia noted, Peripheral blood Hgb 11 g/dL, Platelets 100x109/L, Neutrophils 1.0x109/L, Blasts 0%. Partial response: All CR criteria if abnormal before treatment except: Bone marrow blasts decreased by 50% over pretreatment but still > 5% , Cellularity and morphology not relevant; Stable disease - Failure to achieve at least PR, but no evidence of progression for > 8 weeks; No Response or Failure - Death during treatment or disease progression characterized by worsening of cytopenias, increase in percentage of bone marrow blasts, or progression to a more advanced MDS French-American-British (FAB) classification subtype than pretreatme
Time Frame: Baseline up to 2 treatment cycles (8 weeks)
Measure: Number; unit: percentage of participants
Groups:
- Azacytidine + GM-CSF: Azacytidine administered intravenously (IV) or subcutaneously (SQ) at starting dose of 40 mg/m^2, daily for 4 days.
  GM-CSF administered IV or subcutaneously at 250 mcg/m^2 one day (the next day) after completion of azacytidine treatment, for 3 consecutive days.
  Each treatment cycle will last at least 4 weeks
  Azacytidine: Starting dose: 40 mg/m^2 intravenously (IV) or subcutaneously (SQ) daily for 4 days.
  GM-CSF: 250 mcg/m^2 IV or SQ one day (the next day) after completion of azacytidine treatment, for 3 consecutive days.
Arm/Group | Azacytidine + GM-CSF
Number analyzed (Participants) | 8
percentage of participants
  Complete Response (CR) | 0
  Partial Response (PR) | 0
  No Response | 100

ADVERSE EVENTS:
Time Frame: Adverse events captured from the time of participant consent until 30 days after the last dose of drug.
Arm/Group | Azacytidine + GM-CSF
Serious Adverse Events (participants affected / at risk) | 3/8
Other Adverse Events (participants affected / at risk) | 8/8
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Azacytidine + GM-CSF (N=8)
Fever (General disorders) | 1 (1)
Injection Site Reaction (Infections and infestations) | 1 (1)
Urinary Tract Infection (Infections and infestations) | 1 (1)
Bone Pain (General disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Azacytidine + GM-CSF (N=8)
Fever (General disorders) | 4 (6)
Nausea/Vomiting (Gastrointestinal disorders) | 4 (6)
Diarrhea (Gastrointestinal disorders) | 2 (3)
Chest Pain (General disorders) | 1 (1)
Consipation (Gastrointestinal disorders) | 3 (3)
Fatigue (General disorders) | 4 (4)
Shortness of Breath (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Dizziness (Nervous system disorders) | 1 (1)
Memory Change (Nervous system disorders) | 1 (3)
Blurred Vision (Nervous system disorders) | 1 (2)
Muscle Pain (General disorders) | 3 (4)
Upper Respiratory Infecion (Infections and infestations) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Mouth Pain (General disorders) | 2 (2)
Bone Pain (General disorders) | 1 (1)
Vertigo (Nervous system disorders) | 1 (1)
Eye Dryness (General disorders) | 1 (2)
Injection Site Reaction (General disorders) | 1 (1)
Verebral Fracture (Musculoskeletal and connective tissue disorders) | 1 (1)
Hypotension (Vascular disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No